CLINICAL TRIAL: NCT04688398
Title: Study of the Impact of Fatty Acids From Seal Oil on the Relief of Symptoms Associated With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Ministry of Agriculture, Fisheries and Food, Quebec (Other Government); Groupe De Recherche En Rhumatologie Et Maladies Osseuses Inc. (Industry)
Responsible Party: Principal Investigator, Alain Doyen, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019101
Record Dates: First submitted 2020-12-14; First posted 2020-12-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Polyarthritis
Keywords: seal oil; inflammation
MeSH Terms: conditions — Arthritis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seal oil (Experimental): Daily intake of 15 ml of seal oil containing 534 mg of EPA + 1129 mg of DHA + 530 mg of DPA during 12 weeks
  Interventions: Dietary Supplement: Seal oil
- Control (Active Comparator): Daily intake of vegetable oil during 12 weeks
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Seal oil — Consumption of seal oil once per day (at breakfast)
  Arms: Seal oil
Dietary Supplement: Control — Consumption of vegetable oil once per day (at breakfast)
  Arms: Control

SUMMARY:
This project proposes to conduct the first fully controlled and randomized clinical study demonstrating the impact of DPA-rich sea bass oil on the reduction of symptoms related to rheumatoid arthritis. This unique approach will allow to clinically evaluate the benefits of sea bass oil on the relief of rheumatoid arthritis-related pain in a population suffering from inflammatory arthritis.

DETAILED DESCRIPTION:
The main objective of this project is to measure the efficacy of DPA-rich marine seal oil in improving the clinical signs and symptoms associated with rheumatoid arthritis through the score calculated from the Rheumatoid Arthritis Disease Activity Index (RADAI) questionnaire, in patients suffering from this disease.

The secondary objectives are to evaluate the effect of DPA-rich seal oil on:

1. the degree of disease activity as measured by a joint examination performed by the physician
2. the patient's overall health, quality of life and level of fatigue
3. blood biomarkers of inflammation (CRP: c-reactive protein, TNF-: tumor necrosis factor, IL-1, IL-6 and IL-17: interleukin);
4. the use of non-steroidal anti-inflammatory drugs (NSAIDs);
5. the occurrence of side effects.

To do so, the proposed study is a multi-center, randomized, double-blind, parallel-designed study involving 130 participants with a previous diagnosis of RA from two research and treatment centers in Quebec: the "Groupe de recherche en rhumatologie et maladies osseuses" (GRMO Inc.) from Québec and the "Centre de recherche musculo-squelettique" (CRMS) from Centre du Québec. Rheumatologists from each of the centers, as well as research nurses, will be involved in this project, which will be coordinated by a research professional from the Institut sur la nutrition et les aliments fonctionnels (INAF) at Université Laval. Half of the participants (n=65) will randomly receive the experimental treatment (marine seal oil) while the other half will receive the control treatment (vegetable oil). In order to reach a minimum blood concentration of omega-3 fatty acids for measurable effects, the experimental and control treatments will be administered over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with RA after the age of 18;
* Have had RA for at least 1 year;
* Meet the 2010 ACR/EULAR criteria;
* Stable disease status for at least 3 months:

  * Low to moderate activity as measured by the Clinical Disease Activity Index (CDAI);
  * Stable dose of DMARD (conventional synthetic Disease Modifying Anti-Rheumatic Drug) for at least 3 months;
  * Stable dose of NSAIDs and corticosteroids for at least 1 month;
  * Do not take > 10 mg per day of prednisone.

Exclusion Criteria:

* Have been diagnosed with another rheumatologic autoimmune disease;
* Have been diagnosed with inflammatory bowel disease (ulcerative colitis or Crohn's disease);
* Have a disease that may interfere with the physician's assessment (e.g. severe osteoarthritis);
* Have fibromyalgia;
* Consume omega-3 fatty acid supplements other than those given during the project;
* Have an allergy or intolerance to seafood;
* Consume natural health products that may potentially affect inflammation (e.g. glucosamine, chondroitin, devil's claw, curcumin products) during the project;
* Consume more than two servings (1 serving = 90 g or 3 ounces) of fish and seafood per week for the duration of the study;
* Take anticoagulant medication;
* Be treated or have previously received biological agents or inhibitors of JAK (Janus kinase) (family of tyrosine kinases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of DPA-rich seal oil in improving the clinical signs and symptoms associated with rheumatoid arthritis | One year after the beginning of the study
  Change in the RADAI (Rheumatoid Arthritis Disease Activity Index) score post intervention is measured with a self-administrated questionnaire of 5 questions. Total score can vary from 0 to 10. Higher the score, higher the signs and symptoms.

SECONDARY OUTCOMES:
Degree of disease activity through the 66/68-swollen and tender joint count (SJC66/TJC68) | One year after the beginning of the study
  Measured by doctor's joint examination on 66/68 joints (number of painful and swollen joints). The 66/68-swollen and tender joint count (SJC66/TJC68) is a common questionnaire used for rheumatoid arthritis. The joints count is scored as a sum of the tender joints and the sum of the swollen joints. Higher the score, higher the disease activity.
Overall blood biomarkers of inflammation (cytokines) | One year after the beginning of the study
  Measured via TNF-alpha, IL-1, IL-6 and IL-17 through a kit.
Overall inflammation | One year after the beginning of the study
  Measured via blood CRP.
Patient's overall health | One year after the beginning of the study
  Measured by a self-administrated questionnaire called Health Assessment Questionnaire (HAQ). Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). Result of this questionnaire is a mean score between 0 to 3. Higher the score, higher the difficulties related to the overall health issues.
Patient's quality of life measured with MOS 36-item short-form health survey (SF36) | One year after the beginning of the study
  Measured by a self-administrated questionnaire called Medical Outcome Study Short Form-36 or MOS 36-item short-form health survey (SF36). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The higher the score the less disability.
Patient's level of fatigue | One year after the beginning of the study
  Measured with the FACIT fatigue-scale (version 4) which is a self-administrated questionnaire. Each of the 13 questions is scaled from 0 to 4. After summing all the items, the total is reported on 100. The higher the score, the better the quality of life.
Change in the use of non-steroidal anti-inflammatory drugs | One year after the beginning of the study
  Self-reported by the participant by filling a daily form reporting the consumption of non-steroidal anti-inflammatory drugs. The use of these drugs during study will be compared to the use of these drugs during the washout phase.
Rate of occurrence of side effects between experimental group and control group. | One year after the beginning of the study
  Self-reported by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Doyen, PhD, Principal Investigator — Laval University
Locations (1):
- GRMO, Québec, Canada